CLINICAL TRIAL: NCT03924973
Title: Long-term Efficacy of Early Intervention With Early Start Denver Model (ESDM) on the Severity of Autism
Brief Title: 3 Year Follow up Study of the IDEA Population
Acronym: IDEA2SCOLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-A02446-47
Record Dates: First submitted 2019-04-19; First posted 2019-04-23 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: single blind
Who Masked: Outcomes Assessor
Masking Description: randomization will follow that of the IDEA study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Children below the age of 3 in this group received 2 years of ESDM intervention for 12 hours per week, and then treatment as usual for the 3 following years.
  What is called "treatment as usual" is what the community can usually offer. That is what the control group in IDEA received.
  In IDEA-2, both control and interventional group of IDEA will receive treatment as usual during 3 years.
  Treatment as usual comprises of different types of interventions, such as speech pathology therapy, occupational therapy and other types of therapy more or less specific to ASD in the community.
  Interventions: Behavioral: ESDM followed by treatment as usual
- Control group (Other): Children in this group received treatment as usual delivered in the community for the 2 years of IDEA.
  Participants will still receive treatment as usual delivered in the community during IDEA-2, in the 3 years following IDEA.
  Interventions: Behavioral: ESDM followed by treatment as usual

INTERVENTIONS:
Behavioral: ESDM followed by treatment as usual — The intervention was ESDM, delivered by professionals, one therapist per child, 12 hours per week during 2 years.
  Then, they will receive the treatment as usual during 3 years in this current follow-up study.
  Precise description of the 2 years ESDM treatment can be found in the published protocol of IDEA.
  What is called "treatment as usual" is what the community can usually offer. That is what the control group in IDEA received.
  In IDEA-2, both control and interventional group of IDEA will receive treatment as usual during 3 years.
  Treatment as usual comprises of different types of interventions, such as speech pathology therapy, occupational therapy and other types of therapy more or less specific to ASD in the community.
  All the interventions received by the children will be monitored in IDEA-2. All different treatment approaches will be quantified (type, frequency, intensity and duration).
  Other Names: Treatment as usual delivered in the community

SUMMARY:
The aim of this study is to assess the efficiency of early treatment for ASD children 5 years after initial treatment.

The early treatment implemented was 12 hours per week of ESDM versus treatment as usual during 2 years. This was done as an RCT, called IDEA. Children will now be included in IDEA-2 SCOLA, a three year follow up study.

DETAILED DESCRIPTION:
180 children with ASD, younger than 3 years old, were included in the IDEA RCT. Children were allocated to the ESDM treatment group or the treatment as usual group. The aim of IDEA-2 is to follow-up this population for 3 years after the initial 2 years of intervention, that is, 5 years after initial inclusion to IDEA.

Investigators hypothesize that children who received ESDM 12 hours per week will have a significant decrease of autism symptoms and will have a better scholastic level 5 years after initial inclusion to IDEA.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in the initial IDEA trail
* Requiring less than 40 minutes travel to the assessment center

Exclusion Criteria:

* Impossibility of coming in for assessment
* Exclusion from IDEA

Ages: 39 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
ADOS (Autism Diagnostic Observation Schedule ) | 3 YEARS
  Autism Diagnostic Observation Schedule is a semi-structured, standardized, observational tool, which measures core autism symptoms, that is to say reciprocal sociocommunicative interaction, and repetitive and restrictive behaviors. This assessment will be administered by an assessor blind to the allocation group.

SECONDARY OUTCOMES:
Wechsler (Wechsler Intelligence Scale for Children) | 3 YEARS
  The WISC-IV, the Wechsler Intelligence Scale for Children and Adolescents - 4th Edition - measures total IQ as well as 4 indices: verbal comprehension, perceptual reasoning, processing speed and working memory. It is for children aged 6 to 16 and lasts 60 to 90 minutes.
  The WPPSI-R or the Revised Wechsler Primary and Preschool Intelligence Scale is a psychometric test for very young children, for children from 2 to 6 years old The scores of standard items are between 7 and 13 for the average, if they are less than 4, the child is very deficient in this item.
  3 years after the beginning of the follow-up study ( i.e. 5 years after initial inclusion to IDEA
VABS (Vineland Adaptive Behavior Scales) | 3 YEARS
  The items refer to the age of the person: the first items correspond to the simplest tasks that even a small child should know how to do, and at the end of the scale are grouped the most complex tasks.
  In the field of communication: items range from 1 to 67.Depending on the standard score obtained, five adaptive levels can be defined:top, moderately High, adequate, moderately low, low Daily adaptive skills measured by the composite score from the Vineland Adaptive Behavior Scales ( VABS) 3 years after the beginning of the follow-up study ( i.e. 5 years after initial inclusion to IDEA
PPVT ( Peabody Picture Vocabulary Test ) | 3 YEARS
  Receptive language skills measured by Peabody Picture Vocabulary Test (PPVT)3 years after the beginning of the follow-up study ( i.e. 5 years after initial inclusion to IDEA
Parental self-assentiment | 3 YEARS
  Scholastic skills and interventions measured by Parental self-assentiment

CONTACTS AND LOCATIONS:
Overall Officials: GEOFFRAY MARIE-MAUDE, PH, Principal Investigator — CH LE VINATIER
Locations (1):
- Hopital Vinatier, Bron, France